CLINICAL TRIAL: NCT06145477
Title: Parenting for Tomorrow: A New Model for Supporting Preschool Children's Mental Health in Head Start
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: The Rita and Alex Hillman Foundation (Unknown); Richman Foundation (Unknown); Sherman Family Foundation (Unknown); Blanket Fort Foundation (Unknown); Wright Family Foundation (Unknown); Abell Foundation (Other); Baltimore Community Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00404061
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Parenting; Parenting Intervention
Keywords: Parenting; Chicago Parent Program; CPPi

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents enroll in Parenting for Tomorrow using Chicago Parent Program - individualized for families: Parents enroll in Parenting for Tomorrow using Chicago Parent Program - individualized for families (CPPi) implemented through a telehealth approach.
  Interventions: Behavioral: Chicago Parent Program - individualized for families (CPPi)

INTERVENTIONS:
Behavioral: Chicago Parent Program - individualized for families (CPPi) — CPPi is a 8-12 session individual- based parenting skills program

SUMMARY:
Purpose of this study is to test the preliminary efficacy, acceptability, accessibility, cost, and sustainability of an innovative mental health treatment model for young children from low-income, under-resourced communities through a partnership with Head Start programs in urban and rural communities in Maryland.

DETAILED DESCRIPTION:
The purpose of the study is to test the preliminary efficacy, acceptability, accessibility, cost, and sustainability of an innovative, scalable model for improving young children's mental health services through a partnership with Head Start programs in urban and rural communities in Maryland. The study will use four transformational innovations for eliminating barriers to high quality mental health services for families of young children (2-5 years old) from low-income, under-resourced communities through a partnership with Head Start programs in urban and rural communities in Maryland: 1) test an adaptation of a validated group-based parenting skills and support program (Chicago Parent Program) developed in collaboration with African American and Hispanic parents from low-income communities, for use with individual families (CPPi) concerned about the participant's preschool children's mental health; 2) embed CPPi in a trusted community-based agency long committed to a 2-generation social service model of supporting families from low-income communities; 3) use human centered design strategies to co-create a CPPi referral and enrollment strategy with parents and staff that is welcoming, culturally appropriate, consistent with Head Start's service delivery processes, and eliminates the stigma associated with children receiving a psychiatric diagnosis (as is typically required for reimbursement in traditional child mental health settings); and 4) capitalize on the knowledge, experience, and holistic orientation of registered nurses (RNs) to implement CPPi in Head Start. Children's behavior problems collected at baseline and post-intervention data from the parent and teacher's perspectives. Parent satisfaction with CPPi is measured at post-intervention only.

ELIGIBILITY:
Inclusion Criteria:

* Child is 2-5 years old, enrolled in Baltimore City Head Start (Baltimore City Mayor's Office on Child & Family Success) or Head Start sites managed by Catholic Charities of MD
* parent expresses concern about the child's behavior or need for parenting support
* parent speaks English or Spanish
* Parent age 18-99 years
* Parent able to participate in virtual intervention sessions

Exclusion Criteria:

* Parent does not speak English or Spanish

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents (defined broadly to include a range of caregivers) of young children (2-5 years old) in Head Start programs in urban and rural communities in Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in Child Social - Emotional and Behavioral Wellbeing as assessed by the Strength & Difficulties Questionnaire (SDQ) | Baseline, immediately after the intervention
  Strength & Difficulties Questionnaire (SDQ), a 25 item measure of children's emotional symptoms (5 items), conduct problems (5 items), hyperactivity/inattention (5 items), peer relationship problems (5 items) and prosocial behavior (5 items). A higher score on the SDQ's emotional symptoms, conduct problems, hyperactivity/inattention, and peer relationship problems scales generally indicates more difficulties in those areas, while a lower score suggests fewer problems. Conversely, a higher score on the prosocial behavior scales indicates more positive social behaviors, while a lower score suggests more difficulties in this area. The score range for total difficulties is 0-40 and the score range for prosocial behavior is 0-10.
Change in Child Anxiety as assessed by the Preschool Anxiety Scale (PAS) | Baseline, immediately after the intervention
  Preschool Anxiety Scale (PAS), a 28-item measure of young children's generalized, social, and separation anxieties; obsessive compulsive disorder, and physical injury fears. The score ranges from 0 - 112. Elevated scores on specific subscales may be indicative of potential concerns in those areas.
Change in Child Social - Emotional and Behavioral Wellbeing in the Classroom as assessed by the Social Competence and Behavior Evaluation (SCBE) | Baseline, immediately after the intervention
  Head Start teacher ratings of children's social competence and behavior in the classroom using the Social Competence and Behavior Evaluation (SCBE), a 30-item measure with 3 subscales measuring children's social competence, anger/aggression, and anxiety/withdrawal. The score ranges from 30-180. A higher score on the social competence subscale suggests that the child displays more positive social behaviors and skills. A higher score on the anger/aggression subscale suggests that the child exhibits more anger and aggressive behaviors. A higher score on the anxiety/withdrawal subscale suggests that the child experiences more anxiety and withdrawal behaviors.
Change in parenting skills as assessed by the Parenting Questionnaire (PQ) | Baseline, immediately after the intervention
  Parenting Questionnaire (PQ) is a validated 40-item measure of parents' use of positive discipline, harsh discipline, and consistency of discipline techniques. The score ranges from 40-200. There are 3 subscales of interest for the parenting questionnaire that include: (1) Warmth: higher scores = greater warmth; (2) Corporal Punishment: higher scores = greater use of corporal punishment, and (3) Following Through on Discipline: higher scores = more likely to follow through on discipline.
Change in parenting confidence as assessed by the Parenting Sense of Competence Scale (PSOC) | Baseline, immediately after the intervention
  Parenting Sense of Competence Scale (PSOC) is a widely used 17-item measure of parents' confidence with managing their child's behavior. The score ranges from 17-102. A higher score indicates a higher parenting sense of competency.
Number of referred children with clinically significant social-emotional and behavioral scores as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will be assessed by collecting information on the number of referred children with clinically significant Social-emotional and behavioral scores. Data will be obtained from CPPi RNs who will document all service encounters.
Length of time (in days) from referral to first CPPi appointment as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the length of time (in days) from referral to first CPPi appointment. Data will be obtained from CPPi RNs who will document all service encounters.
Number of referred families who initiate CPPi treatment as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the number of referred families who initiate CPPi treatment. Data will be obtained from CPPi RNs who will document all service encounters.
Average attendance by parents to scheduled CPPi sessions as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on average attendance by parents to scheduled CPPi sessions. CPPi includes 6 required and 2 optional modules, and parents are expected to attend 8-12 1-hour sessions to complete CPPi. Data will be obtained from CPPi RNs who will document all service encounters.
Number of CPPi modules completed as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the number of CPPi modules completed. CPPi includes 6 required and 2 optional modules. CPPi includes 6 required and 2 optional modules. Data will be obtained from CPPi RNs who will document all service encounters.
Number of parents completing CPPi as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the number of parents completing CPPi. CPPi includes 6 required and 2 optional modules. Data will be obtained from CPPi RNs who will document all service encounters.
Number of missed appointments without cancellation for CPPi sessions as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the number of missed appointments without cancellation for CPPi sessions. Data will be obtained from CPPi RNs who will document all service encounters.
Number of internet connectivity issues experienced during CPPi sessions as assessed by a survey developed by the study team | Immediately after the intervention
  CPPi accessibility will also be assessed by collecting information on the number of internet connectivity issues experienced. Data will be obtained from CPPi RNs who will document all service encounters.
Percentage of improvement in participants' perceived effectiveness of CPPi as assessed by a survey developed by the study team | Immediately after the intervention
  The CPPi acceptability will be assessed by measuring the impact of CPPi on participants' perceived efficacy.
Percentage of participants reporting satisfaction with the CPPi referral, scheduling process, and virtual format as assessed by a survey developed by the study team. | Immediately after the intervention
  The CPPi acceptability will also be assessed by measuring the referral, scheduling process, and virtual format for CPPi sessions.
Percentage of participants rating CPPi as user-friendly as assessed by a survey developed by the study team. | Immediately after the intervention
  The CPPi acceptability will also be assessed by measuring the ease of use of the intervention program. Data will be collected from parents and RNs who were involved in the program.
Participants' ratings of the quality of therapeutic relationship with CPPi nurses as assessed by a survey developed by the study team. | Immediately after the intervention
  The CPPi acceptability will also be assessed by measuring the quality of therapeutic relationship between parents and the CPPi nurses.
Parent's satisfaction as assessed by a survey developed by the study team | Immediately after the intervention
  Parent's satisfaction will be measured using the Chicago Parent Program Parent Satisfaction Form. Measure includes 19 items assessing the extent to which they and their child benefitted from the program (scored on a Likert-type scale), aspects of the program that were most and least beneficial, and the extent to which they would recommend the program to other parents. Each item is scored and interpreted separately. The score for the first seven questions ranges from 7-28, with a higher score indicating higher satisfaction with the program. For question number 10-16, the score ranges from 7-28, and higher score indicates that the program was very helpful.
CPPi sustainability as assessed by a survey developed by the study team | Immediately after the intervention
  The CPPi sustainability will be measured using interviews that will be conducted with Head Start teachers, family service workers, and agency leaders (n=20) to learn their perceptions of the benefits and limitations of implementing CPPi with their families, extent to which they believe CPPi improved child mental health and contributed to their mission, anticipated barriers and facilitators to sustaining CPPi, and recommendations for future implementation. We will also interview up to 5 CPPi Registered Nurses to learn their perceptions of how CPPi and working with Head Start parents fit with their knowledge, expertise, and career goals and barriers and facilitators to continuing this work after the study ends.
Implementation cost as assessed by a survey developed by the study team | Immediately after the intervention
  The study will estimate CPPi implementation costs including direct (CPPi materials, provider training, referral costs, RN time to prepare for and implement CPPi sessions, RN supervision costs, costs to parents and RN's associated with use of their computer hardware or cellphone and broadband connection, technical problems resulting in additional costs) and indirect (e.g., parent time) costs. Data will come from study records and participant interviews. Costs will be calculated by multiplying the quantity of each source used by the resource's cost per unit, then summing up all of the resources. Person time costs will be estimated using national US Bureau of Labor Statistics mean hourly compensation cost estimates for RNs including salary and fringe benefits. Costs for use of computer equipment and broadband will be estimated based on national average broadband costs per hour allocated to each CPPi participant and RN proportionally based on time in sessions.
Percent of CPPi nurses who adhere to the CPPi program as assessed by a survey developed by the study team | Immediately after the intervention
  All CPPi sessions will be audio recorded (with parent consent) and submitted to the Project Director. A random selection of 10% of audio recordings will be assessed for CPPi Fidelity (RN adherence to the CPPi protocol and facilitation skill/quality).
Number of CPPi sessions attended by the parents as assessed by a survey developed by the study team | Immediately after the intervention
  The CPPi Program participation ranges from 0-12 sessions.

SECONDARY OUTCOMES:
Change in parental mental health - anxiety as assessed by the Generalized Anxiety Disorder Scale (GAD-7) | Baseline, immediately after the intervention
  Generalized Anxiety Disorder Scale (GAD-7) is a 7-item screening measure of generalized anxiety. The score ranges from 0-21. A score of 0-4: indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety.
Change in parental mental health - depressive symptoms as assessed by the Patient Health Questionnaire-Depression Scale (PHQ-8) | Baseline, immediately after the intervention
  Patient Health Questionnaire-Depression Scale (PHQ-8) is a brief measure of depressive symptoms in the general population. The score ranges 0-24. A score of 10 or greater is considered major depression, 20 or more is severe major depression.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gross, DNSc, Principal Investigator — JHU School Of Nursing
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States